CLINICAL TRIAL: NCT01648790
Title: Relative Bioavailability of Prasugrel Orally Disintegrating Tablet Formulations and the Effect of Food on the Bioavailability of the Orally Disintegrating Tablet in Healthy Subjects
Brief Title: A Study of Prasugrel in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 14686; H7T-EW-TAEQ (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-07-20; First posted 2012-07-24 (Estimated); Results first posted 2013-11-05 (Estimated); Last update posted 2013-11-05 (Estimated); Status verified 2013-08

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Prasugrel Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- 5 mg Prasugrel (ODT1) (Experimental): 5 mg Prasugrel as orally disintegrating tablet without Magnasweet® (ODT1) formulation administered once in the fasted state.
  Interventions: Drug: Prasugrel ODT1 - Tablet
- 5 mg Prasugrel (ODT2) (Experimental): 5 mg Prasugrel as orally disintegrating tablet containing Magnasweet® (ODT2) formulation administered once in the fasted state.
  Interventions: Drug: Prasugrel ODT2 - Tablet
- 5 mg Prasugrel (ODT2)-Suspension (Experimental): 5 mg Prasugrel as ODT2 formulation dispersed in water administered once, in the fasted state.
  Interventions: Drug: Prasugrel ODT2 - Suspension
- 5 mg Prasugrel (ODT2)-Fed (Experimental): 5 mg Prasugrel as ODT2 formulation administered once, following a standardized breakfast.
  Interventions: Drug: Prasugrel ODT2 - Tablet
- 2 mg Prasugrel (ODT2) (Experimental): 2 mg Prasugrel as ODT2 formulation administered once in the fasted state.
  Interventions: Drug: Prasugrel ODT2 - Tablet

INTERVENTIONS:
Drug: Prasugrel ODT1 - Tablet — Administered orally as tablet.
  Other Names: LY640315; Effient; Efient
  Arms: 5 mg Prasugrel (ODT1)
Drug: Prasugrel ODT2 - Tablet — Administered orally as tablet.
  Other Names: LY640315; Effient; Efient
  Arms: 2 mg Prasugrel (ODT2); 5 mg Prasugrel (ODT2); 5 mg Prasugrel (ODT2)-Fed
Drug: Prasugrel ODT2 - Suspension — Administered orally as suspension.
  Other Names: LY640315; Effient; Efient
  Arms: 5 mg Prasugrel (ODT2)-Suspension

SUMMARY:
The purpose of this study is to evaluate the amount of drug available in the body when given to healthy participants as two different formulations with or without a meal. In addition, this study will evaluate how much of the drug gets into the blood stream and how long the body takes to get rid of it. Information about any side effects that may occur will also be collected. Each participant will receive a total of five different treatments. Each treatment is given by mouth, once a day. The treatment period lasts for five consecutive days.

DETAILED DESCRIPTION:
The reference formulation is an orally disintegrating tablet without Magnasweet® (ODT1) and the test formulation is an orally disintegrating tablet containing Magnasweet® (ODT2).

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) of 18.5 to 32.0 kilograms per square meter (kg/m^2)

Exclusion Criteria:

* No known allergies to Prasugrel or related compound
* No regular alcohol intake greater than 21 units per week for males or 14 units per week for females

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-07; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were to be given 5 single doses of prasugrel in 5 different sequences on each of 5 consecutive mornings of treatment.
Groups:
- Sequence 1: Day 1= 5 milligrams (mg) prasugrel without Magnasweet (reference) orally disintegrating tablet (ODT1), given on top of tongue in fasted state (T-Fast); Day 2= 5 mg prasugrel with Magnasweet (test) orally disintegrating tablet (ODT2),T-Fast; Day 3= 5 mg test ODT2, given dispersed in water in fasted state (W-Fast); Day 4= 5 mg test ODT2, given on top of tongue in fed state (T-Fed); Day 5= 2 mg test ODT2, T-Fast
- Sequence 2: Day 1= 2 mg test ODT2, T-Fast; Day 2= 5 mg ODT1, T-Fast; Day 3= 5 mg test ODT2, T-Fast; Day 4= 5 mg test ODT2, W-Fast; Day 5= 5 mg test ODT2, T-Fed
- Sequence 3: Day 1= 5 mg test ODT2, T-Fed; Day 2= 2 mg test ODT2, T-Fast; Day 3= 5 mg ODT1, T-Fast; Day 4= 5 mg test ODT2, T-Fast; Day 5= 5 mg test ODT2, W-Fast
- Sequence 4: Day 1= 5 mg test ODT2, W-Fast; Day 2= 5 mg test ODT2, T-Fed; Day 3= 2 mg test ODT2, T-Fast; Day 4= 5 mg ODT1,T-Fast; Day 5= 5 mg test ODT2, T-Fast
- Sequence 5: Day 1= 5 mg test ODT2, T-Fast; Day 2= 5 mg test ODT2, W-Fast; Day 3= 5 mg test ODT2, T-Fed; Day 4= 2 mg test ODT2, T-Fast; Day 5= 5 mg ODT1, T-Fast
Period: Treatment 1
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5
Started | 4 | 4 | 4 | 4 | 4
Received at Least 1 Dose of Study Drug | 4 | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Treatment 2
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5
Started | 4 | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Treatment 3
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5
Started | 4 | 4 | 4 | 4 (Withdrew consent prior to dosing on this treatment day.) | 4
Completed | 4 | 4 | 4 | 3 | 4
Not Completed | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0
Period: Treatment 4
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5
Started | 4 | 4 | 4 | 3 | 4
Completed | 4 | 4 | 4 | 3 | 4
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Treatment 5
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5
Started | 4 | 4 | 4 | 3 | 4
Completed | 4 | 4 | 4 | 3 | 4
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: 5 mg Prasugrel as orally disintegrating tablet without Magnasweet® formulation (ODT1) or orally disintegrating tablet containing Magnasweet® formulation (ODT2) given either on top of tongue or dispersed in water administered in either the fasted or fed state. 2 mg prasugrel ODT2 given on top of tongue in the fasted state.
Arm/Group | All Participants
Number analyzed (Participants) | 20
Age Continuous [Mean (Standard Deviation); unit: years] | 39.3 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 11
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics: Maximum Concentration (Cmax) of Prasugrel Test and Reference Formulation
Description: Cmax= maximum concentration measured from predose through 8 hours postdose. Test formulation is defined as the orally disintegrating tablet containing Magnasweet® (ODT2) and the reference formulation is defined as the orally disintegrating tablet without Magnasweet® (ODT1) specific to the 5 milligrams (mg) prasugrel dosing. Pharmacokinetics will measure prasugrel's (LY640315) active metabolite.
Time Frame: Predose through 8 Hours Post Dose
Population: Pharmacokinetic population consists of all participants who received at least one dose of study drug and have evaluable pharmacokinetic data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Groups:
- 5 mg Prasugrel (ODT1): 5 mg Prasugrel as orally disintegrating tablet without Magnasweet® (ODT1) formulation administered orally once in the fasted state.
- 5 mg Prasugrel (ODT2): 5 mg Prasugrel as orally disintegrating tablet containing Magnasweet® (ODT2) formulation administered orally once in the fasted state.
Arm/Group | 5 mg Prasugrel (ODT1) | 5 mg Prasugrel (ODT2)
Number analyzed (Participants) | 19 | 19
nanograms per milliliter (ng/mL) | 28.6 (41) | 28.1 (51)
Statistical Analysis 1: Comparison: 5 mg Prasugrel (ODT1) vs 5 mg Prasugrel (ODT2); Test type: Superiority or Other; Ratio of Geometric Least Squares Means = 0.983, 90% CI 2-sided [0.819 to 1.18] — Least Squares (LS) means were determined by mixed-effect linear models with treatment, period, sequence as fixed effects, and participants nested within sequence as random effect

2. Primary Outcome: Pharmacokinetics: Area Under the Concentration Curve (AUC) of Prasugrel Reference and Test Formulation
Description: AUC(0-tlast) = area under the concentration versus time curve from time zero to time t, where t is the last time point with a measurable concentration. Test formulation is defined as the orally disintegrating tablet containing Magnasweet® (ODT2) and the reference formulation is defined as the orally disintegrating tablet without Magnasweet® (ODT1) specific to the 5 mg prasugrel dosing. Pharmacokinetics will measure prasugrel's active metabolite.
Time Frame: Predose through 8 Hours Post Dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour per milliliter (ng*h/mL)
Arm/Group | 5 mg Prasugrel (ODT1) | 5 mg Prasugrel (ODT2)
Number analyzed (Participants) | 19 | 19
nanograms*hour per milliliter (ng*h/mL) | 27.1 (31) | 26.8 (38)
Statistical Analysis 1: Comparison: 5 mg Prasugrel (ODT1) vs 5 mg Prasugrel (ODT2); Test type: Superiority or Other; Ratio of Geometric Least Squares Means = 0.987, 90% CI 2-sided [0.918 to 1.06] — LS means were determined by mixed-effect linear models with treatment, period, sequence as fixed effects, and participants nested within sequence as random effect

3. Secondary Outcome: Pharmacokinetics: Maximum Concentration (Cmax) of Prasugrel Test Formulation in Fasted and Fed State
Description: Cmax= maximum concentration measured from predose through 8 hours postdose. Test formulation is defined as the orally disintegrating tablet containing Magnasweet® (ODT2) specific to the 5 mg prasugrel dosing in the fasted and fed state. Pharmacokinetics will measure prasugrel's active metabolite.
Time Frame: Predose through 8 Hours Post Dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Groups:
- 5 mg Prasugrel (ODT2)-Suspension: 5 mg Prasugrel as ODT2 formulation dispersed in water administered once, orally as suspension, in the fasted state.
- 5 mg Prasugrel (ODT2)-Fed: 5 mg Prasugrel as ODT2 formulation administered orally once, following a standardized breakfast.
- 2 mg Prasugrel (ODT2): 2 mg Prasugrel as ODT2 formulation administered orally once in the fasted state.
Arm/Group | 5 mg Prasugrel (ODT1) | 5 mg Prasugrel (ODT2) | 5 mg Prasugrel (ODT2)-Suspension | 5 mg Prasugrel (ODT2)-Fed | 2 mg Prasugrel (ODT2)
Number analyzed (Participants) | 19 | 19 | 20 | 20 | 19
nanograms per milliliter (ng/mL) | 28.6 (41) | 28.1 (51) | 31.5 (45) | 7.79 (60) | 8.81 (47)
Statistical Analysis 1: Comparison: 5 mg Prasugrel (ODT2) vs 5 mg Prasugrel (ODT2)-Fed; Test type: Superiority or Other; Ratio of Geometric Least Squares Means = 0.280, 90% CI 2-sided [0.233 to 0.335] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Pharmacokinetics: Area Under the Concentration Curve (AUC) of Prasugrel Test Formulation in Fasted and Fed State
Description: AUC(0-tlast) = area under the concentration versus time curve from time zero to time t, where t is the last time point with a measurable concentration. Test formulation is defined as the orally disintegrating tablet containing Magnasweet® (ODT2) specific to the 5 mg prasugrel dosing in the fasted and fed state. Pharmacokinetics will measure prasugrel's active metabolite.
Time Frame: Predose through 8 Hours Post Dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour per milliliter (ng*h/mL)
Arm/Group | 5 mg Prasugrel (ODT1) | 5 mg Prasugrel (ODT2) | 5 mg Prasugrel (ODT2)-Suspension | 5 mg Prasugrel (ODT2)-Fed | 2 mg Prasugrel (ODT2)
Number analyzed (Participants) | 19 | 19 | 20 | 20 | 19
nanograms*hour per milliliter (ng*h/mL) | 27.1 (31) | 26.8 (38) | 27 (32) | 20.8 (39) | 8.97 (31)
Statistical Analysis 1: Comparison: 5 mg Prasugrel (ODT2) vs 5 mg Prasugrel (ODT2)-Fed; Test type: Superiority or Other; Ratio of Geometric Least Squares Means = 0.779, 90% CI 2-sided [0.724 to 0.837] — [estimate comment as in outcome 2, analysis 1]

ADVERSE EVENTS:
Arm/Group | 5 mg Prasugrel (ODT1) | 5 mg Prasugrel (ODT2) | 5 mg Prasugrel (ODT2)-Suspension | 5 mg Prasugrel (ODT2)-Fed | 2 mg Prasugrel (ODT2)
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19 | 0/20 | 0/20 | 0/19
Other Adverse Events (participants affected / at risk) | 1/19 | 0/19 | 0/20 | 2/20 | 1/19
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5 mg Prasugrel (ODT1) (N=19) | 5 mg Prasugrel (ODT2) (N=19) | 5 mg Prasugrel (ODT2)-Suspension (N=20) | 5 mg Prasugrel (ODT2)-Fed (N=20) | 2 mg Prasugrel (ODT2) (N=19)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Procedural dizziness (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days